CLINICAL TRIAL: NCT01419080
Title: Patient-centered Outcomes Related to TReatment Practices in Peripheral Arterial Disease: Investigating Trajectories (PORTRAIT Registry)
Brief Title: Patient-centered Outcomes Related to TReatment Practices in Peripheral Arterial Disease: Investigating Trajectories (PORTRAIT)
Acronym: PORTRAIT
Status: Completed | Type: Observational
Sponsor: Saint Luke's Health System (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 11-533
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Peripheral Arterial Disease; Quality of Life; Quality of Care
Keywords: Peripheral Arterial Disease; Quality of Life; Quality of Care
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Peripheral Arterial Disease (PAD) patients: Patients with new onset or exacerbation of peripheral artery (PA) symptoms.

SUMMARY:
An estimated 8 million individuals in America are affected by peripheral arterial disease (PAD), blockages of the leg arteries that can cause excruciating calf pain when walking. PAD can have a tremendous impact on patients' quality of life. It is also associated with high rates of heart attacks and premature death. While there are a number of treatments, there have been few previous studies that have prospectively examined treatment patterns for PAD or sought to systematically identify opportunities to improve care. Most importantly, there have been no rigorous studies examining the impact of the disease from patients' perspectives - their symptoms, function and quality of life - as a function of different patient characteristics and treatments. The PORTRAIT study (Phase II) will systematically document the treatments and health status (symptom, function and quality of life) outcomes of 840 US patients over the course of one year (assessments at baseline, 3, 6, and 12 months) from 10 centers to address these gaps in knowledge. It will illuminate whether disparities in treatment or health status outcomes exist as a function of patients' age, gender, race, socioeconomic or psychological characteristics. PORTRAIT will substantially elevate the field and identify critical gaps in the way PAD is currently managed, including potential disparities in care, so that the quality of care can be improved.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is a highly prevalent, but undertreated atherosclerotic disease with a disproportionately poor cardiovascular prognosis, as compared with other cardiovascular diseases. Cardiac events are, however, only one manifestation of PAD. Patients' health status (symptoms, function, and quality of life) are critical outcomes from patients' perspectives. To date, there have been no systematic prospective evaluations of disease-specific health status outcomes in PAD and how these vary by treatment and patient characteristics. The long-term goal of our work is to create an evidence-based multi-modal PAD management program that can be individualized to each patient. Following our preparatory work in Pilot PCORI grant 1 IP2 PI000753-01, the current proposal will develop a multi-center observational registry called PORTRAIT (Patient-centered Outcomes Related to Treatment Practices in peripheral Arterial disease: Investigating Trajectories). PORTRAIT will prospectively define and relate patients' care to their health status outcomes as a function of their treatment received at specialty clinics for new-onset, or exacerbations, of their PAD. We hypothesize that there will be substantial variability in treatment patterns across providers and by patient characteristics and that these will explain much of the variation in patients' health status outcomes. Four hypothesis-driven specific aims will be tested; the 5th aim will result in a direct deliverable from this study:

Aim 1: We hypothesize strong associations between the severity of patients' health status and the use of revascularization and that these will vary by age, gender, race, and socio-economic status. This aim will examine variations in treatment by patient characteristics as a foundation for identifying disparities in care.

Aim 2: We hypothesize that revascularization will be associated with more rapid, and larger, improvements in health status as compared with non-invasive options, and that these benefits will vary by age, gender, baseline health status, smoking cessation, minority race, and depressive symptoms. The primary objective of PORTRAIT is to quantify patients' PAD-specific health status outcomes overall, and as a function of treatment and patient characteristics.

Aim 3: We hypothesize that variations in performance measure adherence exist across providers, with greater adherence to pharmacologic therapies for prevention, than exercise treatments to improve function. We will compare real world PAD care against 4 PAD performance measures to provide insights into the quality of PAD care.

Aim 4: We hypothesize that variations in pharmacologic and supervised exercise will be associated with differences in health status outcomes and provide the evidence to suggest that failure to prescribe these evidence-based treatments will result in lower health status scores.

Aim 5: Use the new information to create educational tools to assist patients in selecting treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years
* New or recent exacerbation of exertional leg symptoms
* Resting ankle-brachial index assessment ≤0.90 or drop in post-exercise ankle pressure ≥20 mmHg

Exclusion Criteria:

* Non-compressible ankle-brachial index (≥1.30)
* Critical limb ischemia
* Lower-limb endovascular or surgical vascular procedure in past year
* Not speaking either English or Spanish
* Hearing impaired
* Unable to provide written informed consent
* Currently a prisoner

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to a PAD specialty clinic with new-onset exertional leg symptoms, or recent exacerbations of symptoms, will be screened for enrollment at 10 specialty PAD clinics. Trained study coordinators will have access to the outpatient clinic's schedule and be able to identify potentially eligible patients a priori so as to review medical records and identify potential patients. The diagnostic enrollment criterion includes a Doppler resting ankle-brachial index (ABI) ≤0.9026 or a significant drop in post-exercise ankle pressure of ≥20 mmHg. Patients will be asked to participate upon first visiting the PAD clinic, before treatment is started.
  Study coordinators at each center will obtain informed consent and perform the baseline interview at the outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 797 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Smolderen, PhD, Principal Investigator — St. Luke's Hospital, Kansas City, Missouri; John A Spertus, MD, MPH, Principal Investigator — St. Luke's Hospital, Kansas City, Missouri
Locations (10):
- United States (10):
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Yale University, New Haven, Connecticut
  - Ochsner Health System, New Orleans, Louisiana
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island

REFERENCES:
- [Background] Steg PG, Bhatt DL, Wilson PW, D'Agostino R Sr, Ohman EM, Rother J, Liau CS, Hirsch AT, Mas JL, Ikeda Y, Pencina MJ, Goto S; REACH Registry Investigators. One-year cardiovascular event rates in outpatients with atherothrombosis. JAMA. 2007 Mar 21;297(11):1197-206. doi: 10.1001/jama.297.11.1197. PMID 17374814
- [Derived] Smolderen KG, Romain G, Gosch K, Arham A, Provance JB, Spertus JA, Poosala AB, Shishehbor MH, Safley D, Scott K, Stone N, Mena-Hurtado C. Patient knowledge and preferences for peripheral artery disease treatment. Vasc Med. 2023 Oct;28(5):397-403. doi: 10.1177/1358863X231181613. Epub 2023 Aug 28. PMID 37638882
- [Derived] Angraal S, Hejjaji V, Tang Y, Gosch KL, Patel MR, Heyligers J, White CJ, Tutein Nolthenius R, Mena-Hurtado C, Aronow HD, Moneta GL, Fitridge R, Soukas PA, Abbott JD, Secemsky EA, Spertus JA, Smolderen KG. One-Year Health Status Outcomes Following Early Invasive and Noninvasive Treatment in Symptomatic Peripheral Artery Disease. Circ Cardiovasc Interv. 2022 Jun;15(6):e011506. doi: 10.1161/CIRCINTERVENTIONS.121.011506. Epub 2022 May 17. PMID 35579010
- [Derived] Scierka LE, Jelani QU, Smolderen KG, Gosch K, Spertus JA, Mena-Hurtado C, Jones P, Dreyer RP. Patient representativeness of a peripheral artery disease cohort in a randomized control trial versus a real-world cohort: The CLEVER trial versus the PORTRAIT registry. Contemp Clin Trials. 2022 Jan;112:106624. doi: 10.1016/j.cct.2021.106624. Epub 2021 Nov 16. PMID 34793986
- [Derived] Jelani QU, Mena-Hurtado C, Gosch K, Mohammed M, Labrosciano C, Regan C, Scierka LE, Spertus JA, Nagpal S, Smolderen KG. Association of sleep apnea with outcomes in peripheral artery disease: Insights from the PORTRAIT study. PLoS One. 2021 Sep 10;16(9):e0256933. doi: 10.1371/journal.pone.0256933. eCollection 2021. PMID 34506511
- [Derived] Peri-Okonny PA, Wang J, Gosch KL, Patel MR, Shishehbor MH, Safley DL, Abbott JD, Aronow HD, Mena-Hurtado C, Jelani QU, Tang Y, Bunte M, Labrosciano C, Beltrame JF, Spertus JA, Smolderen KG. Establishing Thresholds for Minimal Clinically Important Differences for the Peripheral Artery Disease Questionnaire. Circ Cardiovasc Qual Outcomes. 2021 May;14(5):e007232. doi: 10.1161/CIRCOUTCOMES.120.007232. Epub 2021 May 5. PMID 33947205
- [Derived] Malik AO, Poghni Peri-Okonny, Gosch K, Thomas MB, Mena-Hurtado C, Hiatt W, Aronow HD, Jones PG, Provance J, Labrosciano C, Jelani QU, Spertus JA, Smolderen KG. Association of perceived stress with health status outcomes in patients with peripheral artery disease. J Psychosom Res. 2021 Jan;140:110313. doi: 10.1016/j.jpsychores.2020.110313. Epub 2020 Nov 24. PMID 33279876
- [Derived] Jelani QU, Mena-Hurtado C, Burg M, Soufer R, Gosch K, Jones PG, Spertus JA, Safdar B, Smolderen KG. Relationship Between Depressive Symptoms and Health Status in Peripheral Artery Disease: Role of Sex Differences. J Am Heart Assoc. 2020 Aug 18;9(16):e014583. doi: 10.1161/JAHA.119.014583. Epub 2020 Aug 12. PMID 32781883
- [Derived] Jelani QU, Smolderen KG, Halpin D, Gosch K, Spertus JA, Iyad Ochoa Chaar C, Tutein Nolthenius RP, Heyligers J, De Vries JP, Mena-Hurtado C. Patient profiles and health status outcomes for peripheral artery disease in high-income countries: a comparison between the USA and The Netherlands. Eur Heart J Qual Care Clin Outcomes. 2021 Sep 16;7(5):505-512. doi: 10.1093/ehjqcco/qcaa052. PMID 32539108
- [Derived] Jelani QU, Jhamnani S, Spatz ES, Spertus J, Smolderen KG, Wang J, Desai NR, Jones P, Gosch K, Shah S, Attaran R, Mena-Hurtado C. Financial barriers in accessing medical care for peripheral artery disease are associated with delay of presentation and adverse health status outcomes in the United States. Vasc Med. 2020 Feb;25(1):13-24. doi: 10.1177/1358863X19872542. Epub 2019 Oct 11. PMID 31603393
- [Derived] Smolderen KG, Gosch K, Patel M, Jones WS, Hirsch AT, Beltrame J, Fitridge R, Shishehbor MH, Denollet J, Vriens P, Heyligers J, Stone MEd N, Aronow H, Abbott JD, Labrosciano C, Tutein-Nolthenius R, A Spertus J. PORTRAIT (Patient-Centered Outcomes Related to Treatment Practices in Peripheral Arterial Disease: Investigating Trajectories): Overview of Design and Rationale of an International Prospective Peripheral Arterial Disease Study. Circ Cardiovasc Qual Outcomes. 2018 Feb;11(2):e003860. doi: 10.1161/CIRCOUTCOMES.117.003860. PMID 29440123

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peripheral Arterial Disease (PAD) Patients
Started | 797
Completed | 666
Not Completed | 131
Not completed — Withdrawal by Subject | 75
Not completed — Death | 30
Not completed — Lost to Follow-up | 23
Not completed — Too Ill | 3

BASELINE CHARACTERISTICS:
Population: Difference in number of patients analyzed due to missing information on treatment status.
Arm/Group | Peripheral Arterial Disease (PAD) Patients
Number analyzed (Participants) | 797
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 334
  Male | 463
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 782
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 577
  Race: Black | 183
  Race: Other | 37
Region of Enrollment [Number; unit: participants]
  United States | 797
Peripheral Artery Questionnaire Summary Score Baseline [Mean (Standard Deviation); unit: units on a scale (0-100)] — Scores on a scale of 0-100, with higher scores representing better health status (0= worst health imaginable, 100= best health imaginable). Subscales are weighed in a standardized scoring algorithm (proprietary). Measures symptoms, symptom stability, and quality of life.
  units on a scale (0-100) | 46.8 (22)

OUTCOME MEASURES:

1. Primary Outcome: Peripheral Artery Disease (PAD) - Specific Health Status
Description: Scores on a scale of 0-100 with higher scores representing better health status (0= worst health imaginable, 100= best health imaginable). Subscales are weighed in a standardized scoring algorithm (proprietary). Measures symptoms, symptom stability, and quality of life.
Time Frame: One Year
Measure: Mean (Standard Deviation); unit: units on a scale of 0-100
Groups:
- Received Invasive Treatment: Received invasive treatment (endovascular, surgical) as a primary treatment strategy (<=3 months following enrollment)
- Did Not Receive Invasive Treatment: Did not receive invasive treatment (endovascular, surgical) as a primary treatment strategy (<=3 months following enrollment)
Arm/Group | Received Invasive Treatment | Did Not Receive Invasive Treatment
Number analyzed (Participants) | 141 | 552
units on a scale of 0-100 | 70.7 (25.4) | 66.9 (25.1)

2. Secondary Outcome: All-cause Mortality
Description: all-cause mortality
Time Frame: One Year
Measure: Count of Participants; unit: Participants
Groups:
- Peripheral Artery Disease (PAD) Patients: Patients with new onset or exacerbation of peripheral artery (PA) symptoms.
Arm/Group | Peripheral Artery Disease (PAD) Patients
Number analyzed (Participants) | 797
Participants | 30

ADVERSE EVENTS:
Arm/Group | Peripheral Arterial Disease (PAD) Patients
Serious Adverse Events (participants affected / at risk) | 30/797
Other Adverse Events (participants affected / at risk) | 0/797
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peripheral Arterial Disease (PAD) Patients (N=797)
All cause mortality (General disorders) | 30 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No